CLINICAL TRIAL: NCT04166578
Title: Comparison of Analgetic Effect of Two Solutions of Intracameral Anesthesia During Cataract Surgery: a Pilot Study
Brief Title: Analgetic Effect of Two Solutions of Intracameral Anesthesia During Cataract Surgery in Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Sponsor
Other Study IDs: 002
Record Dates: First submitted 2019-08-13; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Cataract; Analgesia; Ophthalmological Disorder
MeSH Terms: conditions — Cataract; Agnosia; Eye Diseases | interventions — Lidocaine; Lens Implantation, Intraocular; Slit Lamp Microscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mydrane group: Patients were randomly selected to the group receiving intracameral 0.2 ml Mydrane (a solution of 1% lidocaine and 0.025% of adrenaline ) during phacoemulsification.
  Interventions: Drug: lignocaine; Procedure: Phacoemulsyfication; Procedure: Intraocular lens implantation; Behavioral: Visual Analog Scale for Pain; Behavioral: Brief Pain Inventory-short form; Diagnostic Test: Best corrected visual acuity measurment; Diagnostic Test: Slit-lamp biomicroscopy
- Reference group: Patients were randomly selected to the group receiving intracameral a combination of intracameral solution of lignocaine 1% and adrenalin 0.025% (0.2 ml) during phacoemulsification.
  Interventions: Drug: lignocaine; Procedure: Phacoemulsyfication; Procedure: Intraocular lens implantation; Behavioral: Visual Analog Scale for Pain; Behavioral: Brief Pain Inventory-short form; Diagnostic Test: Best corrected visual acuity measurment; Diagnostic Test: Slit-lamp biomicroscopy

INTERVENTIONS:
Drug: lignocaine — The group of 62 patients undergoing cataract surgery received Mydrane (Mydrane group) or a combination of 1% solution of lignocaine and 0.025% solution of adrenalin (reference group) as an intraocular anesthetic
Procedure: Phacoemulsyfication — Phacoemulsification is a technic of cataract surgery in which the eye's internal lens is emulsified with an ultrasonic handpiece and aspirated from the eye.
Procedure: Intraocular lens implantation — An intraocular lens implant is a synthetic, artificial lens placed inside the eye that replaces the focusing power of a natural lens that is surgically removed, usually as part of cataract surgery.
Behavioral: Visual Analog Scale for Pain — VAS for Pain is a new tool developed to assess the pain in quantitative terms.
  Other Names: VAS for pain
Behavioral: Brief Pain Inventory-short form — BPI short form is a tool developed to assess the pain in quantitative terms. The BPI allows patients to rate the severity of the pain and the grade to which their pain interferes with common dimensions of feeling and function.
  Other Names: BPI short form
Diagnostic Test: Best corrected visual acuity measurment — Measurement of the best vision correction that can be achieved, such as glasses, as measured on the standard Snellen eye chart. For example, if your uncorrected eyesight is 20/200, but you can see 20/20 with glasses, your BCVA is 20/20.
  Other Names: BCVA
Diagnostic Test: Slit-lamp biomicroscopy — Slit-lamp biomicroscopy allows study of ocular structures and their relationships.

SUMMARY:
Purpose: The aim of the study was to compare the analgetic effect of two solutions of intracameral anesthesia in patients undergoing cataract surgery and assess the factors influencing the patients' postoperative activities.

Methods: In this prospective, single-blind, randomized study, a group of 62 patients undergoing cataract surgery received Mydrane (Mydrane group) or a combination of 1% solution of lignocaine and 0.025% solution of adrenalin (reference group) as an intraocular anesthetic. The analgetic effect of these two anesthetic methods was evaluated using psychological tools - Visual Analog Scale for Pain (VAS Pain) and Brief Pain Inventory-short form (BPI) on the next day after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* best corrected visual acuity (BCVA) of 0.2 logMAR or worse
* and agreement for taking part in the study

Exclusion Criteria:

* depressive disorder or expected compliance problems (known psychiatric disease)
* epilepsy
* ongoing treatment with hypnotics or psychotropic drugs (including opioids) within a week before admission
* daily analgesic treatment
* intake of additional rescue medications due to the pain after surgery
* omitting postoperative visit
* no consent to complete the survey
* The patients who later needed additional medications for pain relief

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 70 patients was initially scheduled to participate in this study. However, 8 patients did not attend the postoperative visits and were excluded. As a result, only 62 patients were included in the analysis. The mean age (±SD) of patients was 73.95 (±7.82) years. Female to male ratio was 55/45 in Mydrane group and 53/47 in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
The mean pain score measured with VAS Pain | preoperatively
  The mean pain score measured with Visual Analog Scale for Pain (equivalent to 10 degrees).O points represented no pain and that the 10 points represented the most intense pain he or she felt throughout the surgical procedure.
The mean pain score measured with VAS Pain | postoperatively (the next day after surgery- 24 hours)
  The mean pain score measured with Visual Analog Scale for Pain (equivalent to 10 degrees).O points represented no pain and that the 10 points represented the most intense pain he or she felt throughout the surgical procedure.
The range of pain was measured on the next day after surgery with BPI-short | the next day after surgery (24 hours)
  The the mean severity score, the pain interference mean score was measured with Brief Pain Inventory-short form (BPI-short form). BPI is one of the most widely used measurement tools for assessing clinical pain. It contains two domains that measure pain intensity (severity) and the impact of pain on functioning (interference). In the current study, BPI was used to evaluate the severity of pain and the impact of pain on daily function in the previous 24 h. The responses were given using an eleven-point numeric rating scale (NRS) scored 0-10, where 0 = best outcome/does not interfere/no pain/complete pain relief and 10 = worst outcome/completely interferes/most pain/no pain relief.

CONTACTS AND LOCATIONS:
Locations (1):
- General Department of Ophthalmology in Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No